CLINICAL TRIAL: NCT00126321
Title: Phase II Study of Cladribine, High-dose Cytarabine and Idarubicin in Patients With Relapsed Acute Myeloid Leukemia
Brief Title: Cladribine, Cytarabine and Idarubicin in Patients With Relapsed Acute Myelocytic Leukemia (AML)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: PD Dr. Marie von Lilienfeld-Toal, University Hospital, Med. Klinik III, Bonn, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAI
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Leukemia, Myelocytic, Acute
Keywords: AML, relapsed; cladribine; chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cladribine — 2-chlorodeoxyadenosine, 2-CdA

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of cladribine, high-dose cytarabine and idarubicin in the treatment of patients with relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
Considerable progress has been made in the induction therapy of acute myeloid leukemia (AML); however, current therapeutic results are still unsatisfactory in those with relapsed disease. The purine nucleoside analogue cladribine (2-chlorodeoxyadenosine, 2-CdA) has been shown to be a safe and active agent in acute myeloid leukemia. Synergistic interaction between cladribine and cytarabine has been demonstrated in preclinical and clinical studies.

The current multicenter phase II study was initiated to evaluate the efficacy and toxicity of cladribine, high-dose cytarabine, and idarubicin in the treatment of patients with relapsed AML. Adult patients of all age groups can be enrolled in the trial, but elderly patients will be treated with a less dose-intensive regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed AML with a remission duration of at least 6 months after first complete remission (CR) or of at least 3 months after second (or higher) CR
* Age >= 18 years
* Life expectancy of at least three months (without consideration of AML and complications)
* Eastern Cooperative Oncology Group (ECOG) 0-2 (without consideration of AML and complications)
* Written informed consent

Exclusion Criteria:

* Prior therapy of AML with cladribine
* Severe, uncontrolled infection at time of inclusion (enrollment is possible after control of infection)
* Cardiac insufficiency grade III or IV New York Heart Association (NYHA)
* Severe renal insufficiency with a clearance of < 30 ml/min (if not due to AML)
* Severe hepatic insufficiency with bilirubin > 3 mg/dl or AST > 200 U/l (if not due to AML)
* Other severe organ impairment grade III or IV World Health Organization (WHO) (if not due to AML or, in the opinion of the investigator, may not interfere with the procedures in the study)
* HIV infection
* Intolerance to study drugs
* Pregnant or breast-feeding women
* Any other malignant disease which will probably affect the course of AML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Toxicity according to National Cancer Institute/Common Toxicity Criteria (NCI/CTC), especially the rate of severe infections and the death rate | continuous
Rate of complete remission

SECONDARY OUTCOMES:
Remission duration
Overall survival
Influence of cytogenetic aberrations on remission rate, duration of remission and overall survival
Course of CD3/CD4+ subpopulation after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marie von Lilienfeld-Toal, MD, Principal Investigator — Medical Clinic & Policlinic III, University Hospital Bonn
Locations (1):
- Medical Clinic & Policlinic III, University Bonn, Bonn, Germany